CLINICAL TRIAL: NCT06973759
Title: Bright Light Therapy for Adolescents With Depression and Eveningness - a Randomized, Placebo-controlled, Assessor-blinded Study
Brief Title: Adjunctive Bright Light Therapy in Adolescents With Depression and Eveningness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Joey WY Chan, Clinical Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024.494-T; 12230316 (Other Grant/Funding Number: Health and Medical Research Fund (HMRF), Food and Health Bureau, Hong Kong)
Record Dates: First submitted 2025-04-23; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Depression, Unipolar
Keywords: Depression; Eveningness; Bright light therapy; Adolescents
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Ultraviolet Therapy

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The subjects will be explained that the study aims to test the efficacy of the different modalities of non-pharmacological treatments for depression including bright light therapy and dim red light, without mentioning which one is the placebo. An independent outcome assessor will be blinded to the treatment allocation throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright light therapy group (Experimental): Blue-enriched white light
  Interventions: Device: Bright light therapy
- Dim red light group (Placebo Comparator): Dim red light
  Interventions: Device: Dim red light

INTERVENTIONS:
Device: Bright light therapy — Exposure to blue-enriched white light for 15-30 minutes a day for 8 weeks
  Arms: Bright light therapy group
Device: Dim red light — Exposure to dim red light for 15-30 minutes a day for 8 weeks.
  Arms: Dim red light group

SUMMARY:
This study examines the efficacy of bright light therapy as a treatment for adolescents diagnosed with unipolar non-seasonal depression who exhibit an evening chronotype.

DETAILED DESCRIPTION:
This randomized, placebo-controlled, assessor-blinded trial aims to evaluate the efficacy of bright light therapy (BLT) as a treatment for adolescents with depression and evening chronotype. Eligible participants will be randomized to receive either BLT or dim red light (placebo) daily for 8 weeks. Depression severity, sleep parameters, and circadian markers will be assessed at baseline, during treatment, post-treatment, and at follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese, aged 12-19 years old;
2. Written informed assent/consent of participation into the study is given by the participant and his/her parent or guardian (for those aged under 18), respectively;
3. Having a DSM-5 diagnosis of unipolar non-seasonal depression as confirmed by the Chinese version of the Kiddie-Schedule for Affective Disorders and Schizophrenia (K-SADS) psychiatric interview, DSM-5 Seasonal specifier, AND having a score on Children's Depression Rating Scale (CDRS-R) at least 40;
4. Being classified as evening chronotype according to the score on the reduced Horne-Östberg Morning-Eveningness Questionnaire (rMEQ), i.e. <12.

Exclusion Criteria:

1. A current diagnosis of substance abuse or dependence; a current or past history of manic or hypomanic episode, schizophrenia spectrum disorders, organic mental disorders, or intellectual disabilities;
2. Having a clinically significant suicidality (presence of suicidal ideation with a plan or an attempt) as assessed by K-SADS;
3. Having been enrolled in any other clinical trial investigational products within one month at the entry of the study;
4. Initiation of or change in antidepressant medication within past 4 weeks;
5. Having been or is currently receiving any structured psychotherapy;
6. With hearing or speech deficit;
7. Night shift worker;
8. Trans-meridian flight across at least two time zones in the past 3 months and during the study;
9. Presence of an eye disease, e.g., retinal blindness, severe cataract, glaucoma.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of depressive symptoms | Soon after the intervention
  Change in the score of the Children's Depression Rating Scale (CDRS-R), which ranges from 17-113, higher score indicates higher severity of depression.

SECONDARY OUTCOMES:
Change of other clinical symptoms | Soon after the intervention
  Change in Beck Depression Inventory (BDI) score, which ranges from 0-63, higher score indicates greater depression severity.
Change of other clinical symptoms | Soon after the intervention
  Change in Pittsburgh Sleep Quality Index (PSQI) score, which ranges from 0-21, higher score indicates poorer sleep quality.
Change of other clinical symptoms | Soon after the intervention
  Change in Behavior Rating Inventory of Executive Function (BRIEF2) score, which will be transformed into T scores (range = 35 to ≥ 90) for interpretion, higher score indicates higher executive functioning.
Change of other clinical symptoms | Soon after the intervention
  Change in KIDCSREEN-27 score, which ranges from 30-135, higher score indicates better life quality and social support.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No